CLINICAL TRIAL: NCT03993522
Title: Exercise in Patients With a Total Coronary Occlusion
Acronym: EChO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study did not complete recruitment in the time given.
Sponsor: University of Hull (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18/SC/0461
Record Dates: First submitted 2019-05-03; First posted 2019-06-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Coronary Occlusion
Keywords: Chronic Total Occlusion (CTO)
MeSH Terms: conditions — Coronary Occlusion | interventions — Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTO Exerciser (Experimental): 2x Symptom limited cardiopulmonary exercise tests
  1x Sub-maximal cardiopulmonary exercise test (20 minutes)
  Interventions: Other: Symptom limited cardiopulmonary exercise test & Sub-maximal cardiopulmonary exercise test

INTERVENTIONS:
Other: Symptom limited cardiopulmonary exercise test & Sub-maximal cardiopulmonary exercise test — Exercise tests on cycle ergometer for the purpose of collecting expired breath gasses
  Other Names: CPET

SUMMARY:
A coronary chronic total occlusion refers to the long term complete blockage of a blood vessel supplying the heart.

Exercise is beneficial for patients with heart problems, including people with narrowed blood vessels. However, exercise has not previously been tested in patients with a completely blocked blood vessel. Therefore, the aim of this study is to evaluate exercise testing in participants with a coronary chronic total occlusion, and to see if the physiological changes that occur are reproducible when participants are re-tested. Secondly, the study will see if sustained exercise is safe in this population.

Participants will make 3 visits to our Laboratory. During the first two visits participants will complete symptom limited exercise tests using a stationary bike for approximately 8-12 minutes. The bikes' resistance will gradually increase until participants choose to stop or the researcher ends the test. Participants will wear a mask that collects exhaled breath for testing, and will be connected to an electrocardiogram (heart trace monitor), and blood pressure cuff for monitoring throughout the test. During visits one and three patients will also have blood taken pre and post exercise. Researchers will analyse how the amount of oxygen consumed with increasing exercise relates to the participants' heart rate. A plateau in these measures would indicate a change in the heart's blood supply resulting in reduced function. The participants' third visit will involve cycling under the same conditions as previous visits. However, during this test participants will be asked to cycle continuously for 20 minutes at a resistance set by the researchers. This level of resistance is determined from the results of the first test, as the point at which changes in blood flow and heart function occurred.

In the last five minutes of the test patients will have an echocardiogram (heart scan), to look at the heart function.

DETAILED DESCRIPTION:
The main purpose of this research will be to investigate whether or not changes in the heart's blood supply and function can be seen in coronary chronic total occlusion patients, by investigating information collected during a cardiopulmonary exercise test. Secondly, can these patients exercise safely at this level for an extended period of time.

The cardiology department at Castle Hill Hospital treats approximately 40 patients each year who have a single chronic total coronary occlusion. Researchers will recruit 12 consecutive patients who have a complete blockage of one of the major blood vessels to the heart. These recruits will be found either when the diagnosis is made (during a coronary angiogram when dye is injected into the heart blood vessels), or from the dedicated departmental database at Castle Hill Hospital. Patients will be identified by a member of their usual clinical team. Potential participants will be given a patient information leaflet, explaining the aims of the research and what the study involves. A minimum of 48 hours later, patients will be given a follow up call by a member of their usual clinical care team.

During this call if patients are interested in participating they will be asked for their verbal consent to be contacted by the research team, and given the opportunity to ask questions about the study. Patients will then be invited to attend Castle Hill Hospital to discuss the trial in more detail. Patients will be given the chance to ask questions and explain any concerns they have about the research. They will also be reminded that inclusion in the research is voluntary, and that they can choose to leave the study at any time. Once informed consent has been obtained by a member of the research team, participants will proceed with the baseline assessment (Visit 1). Questions will then be asked about their previous medical history, current condition, and medications they are taking. Basic information will also be collected from the participants; such as height, weight, resting heart rate, blood pressure, ECG, (to measure the electrical activity of the heart), echocardiogram (ultrasound imaging of the hearts function, involving gel being placed on the chest and a hand-held device pressed to the area), and a pre-test blood sample. Following these measures, the participant will be asked to ride a stationary bike against increasing resistance until they can no longer continue (approx. 8-12 minutes). During this exercise they will have their exhaled air (collected via mask), heart rate, blood pressure, and electrocardiogram measured throughout. After completing the test a final blood sample will be collected.

After a minimum of 72 hours and a maximum of 2 weeks, participants will be invited back for visit 2. This visit will include a brief health assessment and will otherwise follow the same structure as the previous visit, minus the blood samples pre and post exercise, and resting echocardiogram (heart scan). The purpose of the second visit is to see if the results of the test are reproducible. The main aim of the test is to see if there is a point that can be identified when the heart is no longer able to work any harder. In healthy individuals, as they cycle harder, the oxygen taken from the lungs with each heartbeat would gradually increase. This would be visible to the researchers in the results of the test. When the body is working hard the heart is forced to work hard too. It does this by increasing its stroke volume, which is the amount of blood it squeezes out to the body with each beat. If the stroke volume increases then the amount of oxygen taken each heart beat will increase. If the participant in the test is a patient with a coronary chronic total occlusion then the research team expect that this will not follow the same path. Under normal conditions like sitting, standing, walking and perhaps light cycling it is possible for this patient's heart to supply enough blood to the muscles. However, because the heart itself is a muscle it too needs more oxygen and therefore more blood if it is going to work harder. As the participant exercises, the heart will try to increase it's stroke volume to supply more oxygen. Unfortunately, because the heart has a blocked vessel it will not receive enough blood to be able to increase its stroke volume. Therefore, the amount of oxygen taken each beat will not increase beyond a certain point, and the researchers should see this as a flattening in the results of the test. The research team will use the data collected from the first and second visit to see if this flattening point exists for each participant. If this point is seen in both tests the researcher will prescribe exercise at this level for the third visit.

A minimum of 72 hours and a maximum of 2 weeks after visit 2, patients will be invited back for their third and final visit. This visit will again begin with a brief health assessment before measures of resting heart rate, blood pressure, electrocardiogram, and a blood sample are collected. Participants will then be asked to pedal a stationary bike this time at a personalised resistance for 20 minutes, whilst exhaled gas, heart rate, blood pressure and electrocardiogram are monitored. During the final 5 minutes of exercise the participant will be given a stress echocardiogram (ultrasound scan of the heart). As in visit 1 a blood sample will be taken from the participant after exercise has been completed.

All visits will occur within the department of Cardiology at Castle Hill Hospital. This is a pilot study and therefore, the number of participants has been determined based on previous experience of performing these tests on patients with non-occlusive coronary disease.

ELIGIBILITY:
Inclusion Criteria:

* Single vessel disease with a chronic total occlusion of the right coronary artery, left anterior descending artery, or left circumflex artery, as identified on coronary angiography performed within the preceding 24 months.
* Willingness to undertake maximal cardiopulmonary exercise test
* Resting systolic blood pressure <180mmHg
* Resting Diastolic blood pressure <100mmHg
* Aged >18yrs
* Normal resting left ventricular function
* Able to provide written informed consent

Exclusion Criteria:

* Significant proximal left main stem stenosis.
* Multi-vessel disease (defined as a diameter stenosis of >50% in another major epicardial coronary vessel)
* Absence of exercise-induced ischaemia evidenced by O2/HR or, ΔVO2/ ΔWR inflection at visit 1 and 2
* O2/HR inflection or, ΔVO2/ ΔWR inflection at a respiratory exchange ratio >1.05
* Change in cardiac medications within previous two weeks
* Unstable angina
* Myocardial infarction within the preceding 6 weeks
* Canadian classification system for angina class IV
* Chronic heart failure
* Significant valvular pathology
* Resting ejection fraction <40%
* Severe orthopaedic limitations
* Past history of Complex arrhythmias
* Atrial fibrillation
* Severe COPD
* Symptoms of intermittent claudication
* Unable to provide written informed consent
* Previous permanent pacemaker implant
* Use of short-term GTN within 30 minutes of exercise testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
intra-patient variability in O2/HR and, ΔO2/ΔWR inflections | 3 weeks
  • To assess the intra-patient variability in the occurrence of the O2/HR and, ΔO2/ΔWR inflection in patients with a CTO during an individualised maximal CPET.
Verification of myocardial dysfunction during inflections via stress echocardiography | 6 weeks
  • To verify that the O2/HR and, ΔO2/ΔWR inflection indicates the onset of exercise induced myocardial dysfunction by visual confirmation of its occurrence using stress-echocardiography

SECONDARY OUTCOMES:
Record any signs of myocardial ischemia, along with adverse and serious adverse events during or following sustained exercise at this intensity | 6 weeks
  • To determine the incidence of myocardial ischemia (as detected during cardiopulmonary exercise test) and/or adverse events during sustained exercise prescribed at an intensity equal to the O2/HR and, ΔO2/ΔWR inflection in patients with a CTO

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hoye, MB, ChB, PhD, Principal Investigator — Hull York Medical School
Locations (1):
- Daisy building Castle Hill Hospital, Hull, Cottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT03993522/Prot_SAP_000.pdf